CLINICAL TRIAL: NCT00174863
Title: Evaluation of Two Doses of SR31747A (75 mg and 125 mg) in Non-Metastatic Androgen-Independent Prostate Cancer. Randomized, Double-Blind, Placebo Controlled Phase II Study
Brief Title: Evaluation of SR 31747A Versus Placebo in Androgen-Independent Non Metastatic Prostate Cancer
Acronym: ODYSSEY
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: ICD Study Director, sanofi-aventis
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: EFC5378
Record Dates: First submitted 2005-09-13; First posted 2005-09-15 (Estimated); Last update posted 2008-12-23 (Estimated); Status verified 2008-12

CONDITIONS: Prostatic Neoplasm
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Who Masked: Participant, Investigator

INTERVENTIONS:
Drug: SR31747A

SUMMARY:
To evaluate the efficacy of SR31747 given at 75 or 125mg per day versus placebo in androgen prostate cancer patient without distant metastases with Time to Clinical progression as main objective and PSA parameters, Tumor response, survival , safety,Tumor-related symptoms deterioration Quality of Life, PK analysis as secondary objectives

ELIGIBILITY:
Inclusion Criteria:

* Prior confirmed histological diagnosis of prostatic carcinoma.
* Rising PSA while receiving hormonal therapy or after surgical castration defined as 2 sequential increases above a previous lowest reference value within the past 12 months; PSA must be at least 4ng/ml at the time of study entry.
* No distant metastases as evidenced by bone scan (+ or - centered X-Ray or MRI), and spiral thoracoabdominopelvic CT scan.
* Effective castration throughout the study. Any prior anti-androgen therapy should be stopped with documented continued elevation of PSA 4 weeks after the cessation of flutamide (6 weeks for bicalutamide).
* Serum testosterone levels < 50ng/dL at the time of progression and throughout the study.
* Age > or = to 18 years.
* Extensive metabolizer by CYP2D6 genotyping.
* Karnofsky Performance Status > or = to 70% and life expectancy > 6 months.
* Adequate hematological, renal and liver function.
* Signed written informed consent

Exclusion Criteria:

* Poor metabolizers by CYP2D6 genotyping.
* Prior palliative radiotherapy or any prior chemotherapy or experimental therapy.
* More than one line of any prior anticancer treatment with estrogen (estrogen or estramustine) if discontinued at least 4 weeks before study entry.
* Concomitant administration of biphosphonate or chronic corticosteroids.
* Presence of progressive symptoms not adequately controlled with non opioid medications
* Concomitant use of medications known to be cytochrome P450 2D6 inhibitors as listed in protocol appendice
* Previous malignancies except if there has been a disease-free interval of at least 5 years and except curatively treated non-melanoma skin cancer
* Other serious illness or medical condition, which would not permit the patient to be managed according to the protocol.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 232 (Actual)
Dates: Start 2003-10; Primary Completion 2006-08 (Actual); Study Completion 2006-08 (Actual)

PRIMARY OUTCOMES:
Time To Clinical Progression assessed by every 4 weeks clinical examination and every 12 weeks radiological examinations (Thoraco-abdominopelvic CT scan ; Bone scan ± centered Bone X-rays, MRI)

SECONDARY OUTCOMES:
Every 4 weeks: Clinical examination (safety, Tumor related symptoms deterioration), PSA level determination (PSA endpoints), EuroQoL instrument (Quality of Life), Laboratory tests (Hematology, Biochemistry), one PK sample
Every 12 weeks: radiological examinations (tumor response),

CONTACTS AND LOCATIONS:
Overall Officials: B. TOMBAL, MD, Study Chair — UCL St Luc, Bruxelles BELGIUM
Locations (13):
- sanofi-aventis Australia & New Zealand administrative office, Macquarie Park, New South Wales, Australia
- Sanofi-Aventis Administrative Office, Diegem, Belgium
- Sanofi-Aventis Administrative Office, Laval, Canada
- Sanofi-Aventis Administrative Office, Santiago, Chile
- Sanofi-Aventis Administrative Office, Prague, Czechia
- Sanofi-Aventis Administrative Office, Paris, France
- Sanofi-Aventis Administrative Office, Milan, Italy
- Sanofi-Aventis Administrative Office, México, Mexico
- Sanofi-Aventis Administrative Office, Gouda, Netherlands
- Sanofi-Aventis Administrative Office, Warsaw, Poland
- Sanofi-Aventis Administrative Office, Porto Salvo, Portugal
- Sanofi-Aventis Administrative Office, Barcelona, Spain
- Sanofi-Aventis Administrative Office, Guilford Surrey, United Kingdom

REFERENCES:
- See also: Related Info — http://www.sanofi-aventis.com